CLINICAL TRIAL: NCT04838834
Title: Monitoring Serologic Response to SARS-COV-2 / Coronavirus Disease 2019 (COVID-19) in Children, Adolescents, and Young Adults Receiving Biologic Therapies (RECONN)
Brief Title: Monitoring Serologic Response to Severe Acute Respiratory Syndrome-2 (SARS-COV-2)/COVID-19 in Children
Acronym: RECONN
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: The Jackson Laboratory (Other); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 20-073
Record Dates: First submitted 2021-02-11; First posted 2021-04-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; SARS-CoV-2; Inflammatory Bowel Diseases
Keywords: COVID-19 Serological Testing
MeSH Terms: conditions — COVID-19; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be collected from participants every 3-4 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Individuals susceptible to SARS-CoV-2 and the illness it causes (COVID-19) are comprised of heterogeneous populations with a large risk spectrum for more severe disease. Pre-existing risk factors for a more severe course include respiratory and cardiovascular disease, morbid obesity, diabetes, underlying kidney or liver disease, and immunocompromised status. Whether children and young adults with inflammatory bowel disease (IBD) or juvenile idiopathic arthritis (JIA) receiving immunomodulating biologic and other therapies which are known to increase risk of viral infection are at increased risk of complications from COVID-19 or post-infectious co-morbidities, including the recently described multi inflammatory syndrome (MISC), is entirely unclear. This research focuses on the heretofore uncharacterized immune response to SARS-CoV-2 infection in children and young adults with IBD or JIA who are receiving maintenance immunosuppressive biologic therapies. Given the large Connecticut based infusion program, in a region of the United States with a recent large outbreak of COVID-19, the investigators have a unique opportunity to address a glaring knowledge gap in this unique pediatric, adolescent, and young adult population. The investigators will longitudinally determine antibody development and durability to SARS-CoV-2 in approximately 450-500 children and young adults with IBD or JIA receiving biologic therapy using a highly sensitive and specific quantitative assay utilizing novel technology. This period will include a return to school or work for many with likely resurgent infections, as well as the possible introduction of anti-SARS CoV-2 vaccines. The specific aim is to study the acute and convalescent antibody responses to SARS-CoV-2 infection in a cohort of children and young adults receiving infusions of biologic therapies for IBD and JIA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 2 to 27 years inclusive
2. Patients receiving biologic infusions for inflammatory or rheumatologic disorders at the Connecticut Children's Infusion Center, at a minimum frequency of 2 infusions over a 4 month period
3. Consent/assent as indicated
4. Have vein access placement as standard of care

Exclusion Criteria:

1. Patient and/or parent/legal guardian refused participation
2. Inability to draw requisite blood sample for serum collection

Ages: 2 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults with inflammatory bowel disease or juvenile idiopathic arthritis receiving treatment with biologic agents at Connecticut Children's Infusion Center
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Presence of anti-SARS-CoV-2 Immunoglobulin G (IgG) | At the time of infusions for up to 2 years

SECONDARY OUTCOMES:
Presence of anti-SARS-CoV-2 IgG neutralizing antibodies | At the time of infusions for up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Hyams, MD, Principal Investigator — Connecticut Children's Medical Ctr
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

REFERENCES:
- [Background] Neurath MF. COVID-19 and immunomodulation in IBD. Gut. 2020 Jul;69(7):1335-1342. doi: 10.1136/gutjnl-2020-321269. Epub 2020 Apr 17. PMID 32303609
- [Background] Brenner EJ, Ungaro RC, Gearry RB, Kaplan GG, Kissous-Hunt M, Lewis JD, Ng SC, Rahier JF, Reinisch W, Ruemmele FM, Steinwurz F, Underwood FE, Zhang X, Colombel JF, Kappelman MD. Corticosteroids, But Not TNF Antagonists, Are Associated With Adverse COVID-19 Outcomes in Patients With Inflammatory Bowel Diseases: Results From an International Registry. Gastroenterology. 2020 Aug;159(2):481-491.e3. doi: 10.1053/j.gastro.2020.05.032. Epub 2020 May 18. PMID 32425234
- [Background] Brenner EJ, Pigneur B, Focht G, Zhang X, Ungaro RC, Colombel JF, Turner D, Kappelman MD, Ruemmele FM. Benign Evolution of SARS-Cov2 Infections in Children With Inflammatory Bowel Disease: Results From Two International Databases. Clin Gastroenterol Hepatol. 2021 Feb;19(2):394-396.e5. doi: 10.1016/j.cgh.2020.10.010. Epub 2020 Oct 12. PMID 33059040
- [Background] Robbiani DF, Gaebler C, Muecksch F, Lorenzi JCC, Wang Z, Cho A, Agudelo M, Barnes CO, Gazumyan A, Finkin S, Hagglof T, Oliveira TY, Viant C, Hurley A, Hoffmann HH, Millard KG, Kost RG, Cipolla M, Gordon K, Bianchini F, Chen ST, Ramos V, Patel R, Dizon J, Shimeliovich I, Mendoza P, Hartweger H, Nogueira L, Pack M, Horowitz J, Schmidt F, Weisblum Y, Michailidis E, Ashbrook AW, Waltari E, Pak JE, Huey-Tubman KE, Koranda N, Hoffman PR, West AP Jr, Rice CM, Hatziioannou T, Bjorkman PJ, Bieniasz PD, Caskey M, Nussenzweig MC. Convergent antibody responses to SARS-CoV-2 in convalescent individuals. Nature. 2020 Aug;584(7821):437-442. doi: 10.1038/s41586-020-2456-9. Epub 2020 Jun 18. PMID 32555388
- [Background] Gaebler C, Wang Z, Lorenzi JCC, Muecksch F, Finkin S, Tokuyama M, Cho A, Jankovic M, Schaefer-Babajew D, Oliveira TY, Cipolla M, Viant C, Barnes CO, Hurley A, Turroja M, Gordon K, Millard KG, Ramos V, Schmidt F, Weisblum Y, Jha D, Tankelevich M, Yee J, Shimeliovich I, Robbiani DF, Zhao Z, Gazumyan A, Hatziioannou T, Bjorkman PJ, Mehandru S, Bieniasz PD, Caskey M, Nussenzweig MC, Hagglof T, Schwartz RE, Bram Y, Martinez-Delgado G, Mendoza P, Breton G, Dizon J, Unson-O'Brien C, Patel R. Evolution of Antibody Immunity to SARS-CoV-2. bioRxiv [Preprint]. 2021 Jan 4:2020.11.03.367391. doi: 10.1101/2020.11.03.367391. PMID 33173867
- [Background] Dittadi R, Afshar H, Carraro P. The early antibody response to SARS-Cov-2 infection. Clin Chem Lab Med. 2020 Sep 25;58(10):e201-e203. doi: 10.1515/cclm-2020-0617. No abstract available. PMID 32639941